CLINICAL TRIAL: NCT00767364
Title: Safety and Immunogenicity of Rotavirus Vaccine (RotaTeq(R)) in Infants With Short Bowel Syndrome: A Pilot Study
Brief Title: Safety and Immunogenicity of Rotavirus Vaccine (RotaTeq(R)) in Infants With Short Bowel Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Michigan (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Corewell Health East (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Eric McGrath, Principle Investigator, Children's Hospital of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Merck IISP #35817
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Short Bowel Syndrome
Keywords: Infant
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infants with bowel resection (Experimental): Infants with bowel resection who will receive the oral rotavirus vaccine, RotaTeq(R).
  Interventions: Biological: Oral, live, pentavalent rotavirus vaccine; RotaTeq(R)
- Healthy Infants (Active Comparator): Healthy infants that are gest. age and age-matched controls within 14 days will be given the oral rotavirus vaccine, RotaTeq(R).
  Interventions: Biological: Oral, live, pentavalent rotavirus vaccine; RotaTeq(R)

INTERVENTIONS:
Biological: Oral, live, pentavalent rotavirus vaccine; RotaTeq(R) — Oral vaccine for prevention of rotavirus infection, 3 dose series
  Other Names: RotaTeq vaccine (Merck and Co.)

SUMMARY:
Rotavirus infection is a common pediatric illness and is the leading cause of severe acute gastroenteritis (vomiting and diarrhea) in infants and young children. Since February of 2006, an oral vaccine to prevent rotavirus has been approved by the Food and Drug Administration (FDA). The company that makes the oral vaccine is Merck and Company. Since the FDA approval, the American Academy of Pediatrics (AAP) and that Advisory Committee on Immunization Practices (ACIP) has recommended the use of this oral vaccine in infants. A previous rotavirus oral vaccine, Rotashield, was removed from the market for concerns that it was causing an increase in a gastrointestinal (GI) disease called intussusception. However, the new rotavirus vaccine was studied by the manufacturer and was not found to cause an increase in the cases of intussusception. Intussusception is a disease in which a portion of the GI tract folds back on itself leading to GI tract obstruction or back-up.

The manufacturer of the vaccine noted on package insert information that the vaccine was not studied, originally, in infants with a history of GI disorders or in infants who have had surgery on their abdomen. Currently, there is no information available in the scientific literature about the use of the oral rotavirus vaccine in infants with GI diseases or those who have had GI surgeries.

The objective of the study is the assessment of safety and tolerability of the oral RotaTeq® vaccine for all infants participating in the study. All infants will be followed for clinical adverse events with active safety surveillance for the first 42 days after each dose and also monthly afterward for a total of 12 months from the first vaccination date. The secondary objective of the study is to quantify the immunologic response will occur in all of the infants in the study. Assessment of percentage of the number of infants who have a good immune response (three-fold rise in IgA titer or greater) to the complete rotavirus vaccine series (three oral vaccines in total) by a blood test to check the rotavirus immunoglobulin A (IgA) level in infants with short bowel syndrome compared to normal infants will occur.

Infants, meeting eligibility criteria and whose parents have signed informed consent will have their study information collected. These infants will be tested for the presence of pre-vaccine anti-rotavirus antibody, IgA levels, as mentioned above. After the blood is obtained, participants will receive their first oral rotavirus vaccine dose between the ages of 6 weeks to 12 weeks of life per package insert information. This oral rotavirus vaccine may be administered with other routine pediatric vaccines at the participant primary care provider's office. The date of the rotavirus vaccine and lot number would be recorded on vaccine administration date cards. Most participants will have their vaccines given through the Infectious Disease clinic staff at the Children's Hospital of Michigan.

Subsequent doses of the oral rotavirus vaccine will be given at a minimal interval between vaccines of four weeks. The third, and final vaccine dose must be given by 32 weeks of life. Any adverse reactions to the vaccine will be reported on the National Vaccine Adverse Event Reporting System and MedWatch forms.

Finally, two weeks after the participants have had all three oral rotavirus vaccine doses, the second and final blood draw will take place for measuring the post-vaccine level of anti-rotavirus antibody, IgA.

Participants in the study will be monitored by telephone contacts on days 7, 14, and 42 after each dose and within 48 to 72 hours of each dose of the rotavirus vaccine regarding any serious adverse events. Each infant will also be assessed in the clinical setting each week after a vaccine dose has been given. As above, parents of participants will be asked to fill out the vaccine report card and record the child's temperature, and any episodes of vomiting, diarrhea, blood in the stools or fussiness for the first seven days. The parents will also be asked to record any other events from day 8 through 42 after each vaccine is administered such as fever, ear infection, runny nose, etc. Afterward, parents will also have monthly phone call safety follow-ups during the 12 month period following the first vaccination. A Data Safety and Monitoring Board will oversee the study and it's progress and will have the ability to vote to stop the study.

ELIGIBILITY:
Inclusion Criteria:

* Only those participants whose parents give full informed consent will be included in the study.
* Infants will be eligible for enrolment in the study arm if they have the diagnosis of short bowel syndrome (SBS) and are between the ages of 6 and 12 weeks of age before the start of the vaccine series.
* SBS infants must also be afebrile,

  * have stable to increasing weight,
  * have stable electrolytes and be clinically stable for home discharge (or already discharged home), as assessed by the infant's primary care physicians, prior to administration of the oral RotaTeq® vaccine.
* Study group infants must have at least 30 cm of residual small intestine with a whole colon and intact ileocecal valve or at least 45 cm of residual small intestine (with or without a whole colon) and without an ileocecal valve to be included in the study based on age-related normal lengths from the literature.
* The SBS infant should be at least 10 days post any gastrointestinal surgery at time of vaccine administration and be between 10- to 12- weeks of chronological age at time of first vaccine administration, and be tolerating at least some oral intake (liquids and/or food). The vaccine will not be given in the neonatal intensive care unit for the purposes of this study, although the risk of shedding is low with RotaTeq® vaccine.
* Infants will be eligible for inclusion in the control arm if they have no underlying chronic gastrointestinal medical conditions (Gastro-esophageal Reflux Disease (GERD), is allowed) and
* are between the ages of 6 and 12 weeks of age before the start of the vaccine series.
* Normal control arm infants will be estimated gestational age- and age-matched within 14 days to study arm participants for more accurate comparison between the immune responses.
* These healthy infants will also receive their first vaccine administration at 10- to 12-weeks of chronological age, when possible, so that the immune responses between the groups will be more comparable.

Exclusion Criteria:

* Infants whose parents do not give full informed consent or whom do not meet inclusion criteria will be excluded from participation.
* Additionally, Infants who have a demonstrated history of hypersensitivity to any vaccine component will be excluded.
* Any infant who develops symptoms associated with hypersensitivity reactions after the first or second dose of the vaccine will also be excluded from the study and any further doses.
* Those infants with documented fever of greater than 100.5 degrees F. or severe illness by the end of their 12th week of life and who have not yet received the vaccine will be excluded.
* Any infant who fails to have blood obtained by the third attempt will be automatically excluded from the study.
* Infants with a history of rotavirus or history of receipt of any rotavirus vaccine will be excluded from the study.
* Those infants diagnosed with a congenital or acquired immunodeficiency or neoplasm will be excluded as will any patient who is potentially immunosuppressed (topical and inhaled corticosteroid use would allow for inclusion).
* Infants who have received immunoglobulins will also be excluded (history of receipt of other blood products is allowed).
* Short bowel infants with diagnosed portal hypertension will be excluded.
* Also, any short bowel syndrome infant who is listed or will likely need liver/bowel transplantation (imminent or evident liver failure due to total parenteral nutrition (TPN)-induced liver injury, a total bilirubin level of >7 mg/dl, or stage 2 liver fibrosis, or only two central venous access sites remain) will be excluded from the study.
* In the short bowel syndrome infants, the principal investigator reserves the right to exclude any infant on the basis of any clinical safety concern, such as a specific additional diagnosis, that exists or develops for the individual infant that may be seen as a potential risk factor for a future adverse event.
* Those infants with household contacts who have immunosuppressive conditions, such as infants residing in a household with an immunocompromised person, including individuals with congenital immunodeficiency, HIV infection, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, generalized malignancy, chronic renal failure, nephritic syndrome, organ or bone marrow transplantation, or with those receiving immunosuppressive chemotherapy including long-term systemic corticosteroids will be excluded from the study.
* Any infant that cannot have adequate follow up for safety by telephone or home visit will be excluded from the study.

Ages: 6 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2009-07; Primary Completion 2012-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J McGrath, MD, Principal Investigator — Children's Hospital of Michigan
Locations (3):
- United States (3):
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan

REFERENCES:
- [Background] Parashar UD, Hummelman EG, Bresee JS, Miller MA, Glass RI. Global illness and deaths caused by rotavirus disease in children. Emerg Infect Dis. 2003 May;9(5):565-72. doi: 10.3201/eid0905.020562. PMID 12737740
- [Background] American Academy of Pediatrics Committee on Infectious Diseases. Prevention of rotavirus disease: guidelines for use of rotavirus vaccine. Pediatrics. 2007 Jan;119(1):171-82. doi: 10.1542/peds.2006-3134. PMID 17200286
- [Background] Wales PW, de Silva N, Kim J, Lecce L, To T, Moore A. Neonatal short bowel syndrome: population-based estimates of incidence and mortality rates. J Pediatr Surg. 2004 May;39(5):690-5. doi: 10.1016/j.jpedsurg.2004.01.036. PMID 15137001
- [Background] Wales PW, de Silva N, Kim JH, Lecce L, Sandhu A, Moore AM. Neonatal short bowel syndrome: a cohort study. J Pediatr Surg. 2005 May;40(5):755-62. doi: 10.1016/j.jpedsurg.2005.01.037. PMID 15937809
- [Background] Grosfeld JL, Rescorla FJ, West KW. Short bowel syndrome in infancy and childhood. Analysis of survival in 60 patients. Am J Surg. 1986 Jan;151(1):41-6. doi: 10.1016/0002-9610(86)90009-7. PMID 3080921
- [Background] Centers for Disease Control and Prevention (CDC). Delayed onset and diminished magnitude of rotavirus activity--United States, November 2007-May 2008. MMWR Morb Mortal Wkly Rep. 2008 Jun 27;57(25):697-700. PMID 18583958
- [Background] Goveia MG, Rodriguez ZM, Dallas MJ, Itzler RF, Boslego JW, Heaton PM, DiNubile MJ; REST Study Team. Safety and efficacy of the pentavalent human-bovine (WC3) reassortant rotavirus vaccine in healthy premature infants. Pediatr Infect Dis J. 2007 Dec;26(12):1099-104. doi: 10.1097/INF.0b013e31814521cb. PMID 18043445
- [Background] Parashar UD, Gibson CJ, Bresee JS, Glass RI. Rotavirus and severe childhood diarrhea. Emerg Infect Dis. 2006 Feb;12(2):304-6. doi: 10.3201/eid1202.050006. PMID 16494759

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infants With Bowel Resection | Healthy Infants
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infants With Bowel Resection | Healthy Infants | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Customized [Mean (Full Range); unit: weeks]
  Gestational Age | 31.2 [30 to 40] | 38.6 [37 to 40] | 34.9 [30 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8
Pre-vaccination serum IgA antirotavirus titer [Number; unit: U/ml]
  Subject 1 | 1.56 | 1.56 | 3.12
  Subject 2 | 1.56 | 1.56 | 3.12
  Subject 3 | 1.56 | 1.56 | 3.12
  Subject 4 | 1.56 | NA — There was no control for study Subject 4 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Subject 5 | 1.56 | NA — There was no control subject for study Subject 5 | NA — Total not calculated because data are not available (NA) in one or more arms.
Rotavirus Anti-Immunoglobulin A (IgA) serum antibody level [Geometric Mean (Full Range); unit: U/ml] | 618.61 [259 to 1018] | 431.02 [272 to 935] | 540 [259 to 1018]

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of the Oral RotaTeq® Vaccine
Description: Adverse events and patient tolerance of vaccine doses 1 - 3 for all infants participating in the study were recorded.
Time Frame: 12 months from the first vaccination date
Measure: Number; unit: Individual Adverse Events
Arm/Group | Infants With Bowel Resection | Healthy Infants
Number analyzed (Participants) | 5 | 3
Individual Adverse Events | 18 | 3

2. Secondary Outcome: Serum Anti-rotavirus IgA Level Post-vaccination
Description: Serum anti-rotavirus IgA level was measured post-vaccination in all subjects
Time Frame: 6 months from the first vaccination date
Measure: Number; unit: U/ml
Arm/Group | Infants With Bowel Resection | Healthy Infants
Number analyzed (Participants) | 5 | 3
U/ml
  Participant 1 | 916.4 [260 to 1018] | 935.6 [272 to 935]
  Participant 2 | 679.5 | 314.1
  Participant 3 | 259.7 | 272.5
  Participant 4 | 1018.8 | NA — There was no available control subject for study participant 4
  Participant 5 | 550.0 | NA — There was no available control subject for study participant 5

ADVERSE EVENTS:
Time Frame: 1 year (12 months) from receipt of the first dose of vaccine.
Description: Participant parents were required to keep a symptoms diary and take their son/daughter temperature daily for the first week. Afterwards, the parent was required only to write any symptoms for 42 days on the same paper after each dose. Month phone call follow ups were made to assure that there were no other Adverse Events (AE)s x 12 months.
Arm/Group | Infants With Bowel Resection | Healthy Infants
Serious Adverse Events (participants affected / at risk) | 4/5 | 0/3
Other Adverse Events (participants affected / at risk) | 5/5 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants With Bowel Resection (N=5) | Healthy Infants (N=3)
Low hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Occurred in 1 participant, resolved
Elevated Bilirubin level (Hepatobiliary disorders) | 1 (1) | 0 (0) — Likely due to Chronic TPN use
Fever, Rule out catheter infection (Infections and infestations) | 2 (3) | 0 (0) — Fever and Central catheter, evaluated as Rule out Sepsis
Central Line Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Positive Central Catheter infection, Treatment required inpatient stay
Bowel obstruction; Hirschsprung enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Due to underlying disease, required inpatient stay
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infants With Bowel Resection (N=5) | Healthy Infants (N=3)
Stomal bleeding - hematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0) — Transient stomal site bleeding
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) — No stomal site
Gastrostomy tube drainage after removal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose Stools (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting with diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Fussiness (General disorders) | 1 (1) | 1 (1)
Fever with upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The small sample size makes generalization of the study data difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No